CLINICAL TRIAL: NCT02735096
Title: Palatal Device Providing In-situ Sensory Feedback for Patients With Vestibular Imbalance
Brief Title: Testing an Intraoral Electronic Balance Aid for Vestibular Imbalance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended at the end of 2016
Sponsor: Innervo Technology LLC (Industry)
Collaborators: University of Missouri-Columbia (Other); Blue Ridge Physical Therapy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ICTP216
Record Dates: First submitted 2016-03-30; First posted 2016-04-12 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2018-03

CONDITIONS: Vestibular Disorder
Keywords: Bilateral Vestibular Hypofunction; Unilateral Vestibular Hypofunction; Imbalance
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vestibular Patients for EquiCue Testing (Experimental): Subjects with vestibular deficiency will try the intraoral electronic balance aid to see whether there is improvement in balance.
  Interventions: Device: EquiCue (Intraoral Electronic Balance Aid)

INTERVENTIONS:
Device: EquiCue (Intraoral Electronic Balance Aid) — When the device is worn, a subject will receive small electrical pulses on roof of the mouth as alternative feedback of head tilting or movement.
  Other Names: EquiCue

SUMMARY:
The human body uses vestibular feedback in coordination with visual and somatosensory information to maintain balance and posture. However, various inner-ear disorders due to aging, drug toxicity, viral infections, and injury, etc., may result in loss of vestibular feedback, which makes it difficult for an individual to maintain balance. This study investigates the use of a hidden and noninvasive balance device EquiCue™ V1 developed by Innervo Technology for vestibular substitution. EquiCue™ V1 is a retainer-like intraoral electronic balance aid entirely worn inside the oral cavity and provides in-situ sensory feedback of head tilting and motion on the roof of the mouth. The feedback is delivered by applying small and controlled electrical pulses at precise locations on the palatal surface according to an encoded pattern. This pilot study is to determine how this alternative sensory feedback on the roof of the mouth can be used to improve balance for patients with vestibular loss.

DETAILED DESCRIPTION:
Background

Vestibular imbalance is prevalent in the United States and around the world. According to NIDCD, 4% (8 million) of American adults report a chronic problem with balance (visit vestibular.org for more information). The leading cause of imbalance is vestibular dysfunction. Various vestibular disorders due to aging, diseases, ototoxicity, and injuries, etc. can cause damage or degradation of the vestibular system, resulting in loss of vestibular feedback. Symptoms associated with vestibular loss include: difficulty maintaining straight posture; stumbling or unable to walk straight; lose balance on uneven surfaces or under dim lighting; floating sensation and tendency to look downward to confirm the location of the ground. Vestibular imbalance greatly increases risk of falling and has such disabling effects ranging from reduced activity levels to total loss of mobility.

Vestibular rehabilitation therapies (VRT) may help vestibular patients to compensate with vision and proprioception. However, such compensation is not adequate because the brain often needs a reliable reference in order to use visual and somatosensory information for perception of self-motion and spatial orientation. Consequently, many patients with vestibular imbalance fail to compensate, especially those with profound vestibular loss. Even those who respond to VRT may experience constant physical and mental stress due to overreliance on vision and proprioception that can be misleading in busy environments.

EquiCue™ Intraoral Balance Aid

The intraoral balance aid EquiCue™ V1 is a hidden and noninvasive balance device that vestibular patients can use in various indoor and outdoor activities. It is a retainer-like device entirely worn inside the oral cavity, with no need of surgical implantation, and can be removed when not in use. The device provides in-situ sensory feedback of head tilt and motion by applying small electrical pulses on the roof of the mouth. By sensing the feedback from the device, an individual with vestibular loss can have better judgment of the tilt and motion of the head and make physical adjustment accordingly for better balance of the body. Since the device does not cause alteration to the appearance of the user, patients may use it in public places such as shopping malls, supermarkets, and metro stations, while offering balance assistance and improved postural stability and gait in these busy environments.

Human Subject Study

The current study is an initial stage of a clinical trial on the use of EquiCue™ for patients with vestibular imbalance. The hypothesis is that EquiCue™ can at least partially substitute the lost vestibular function and therefore helps a vestibular patient to achieve better postural stability in daily activities. The basic questions regarding the technology are: 1) How to represent head movement using electrical pulses on the palate; 2) Whether the electrotactile presentation on the palate can be reliably recognized and used for balance control. The study also helps to understand the role of multisensory integration on balance, especially the impact of alternative sensory feedback on the balance system.

Subjects participating in the study will be expected to wear a custom-made retainer-like device and perform movements to test their balance. If a patient is determined to be a suitable subject, the sensitivity profile on the palate of the patient will be measured. After an EquiCue™ intraoral device is custom made, the patient will be asked to fit the device inside the mouth, and verify the basic functionality of the device by identifying direction, perceived intensity, and sensory characteristics of stimuli from the device. The subject will then go through 3-4 sessions of training and testing in which the subject tries to associate the feedback with head movement and to integrate the feedback with other senses to achieve a better spatial orientation and balance. The improvement in balance and gait with the device will be evaluated by using standard tests on balance platforms (Computerized Dynamic Posturography) and Dynamic Gait Index. Tests will be made without wearing the device at the beginning and wearing the device at the end of each training session.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking adults with ages between 18-85.
2. Patients with imbalance resulted from vestibular loss or vestibulopathy.
3. Priority given to those who took vestibular rehabilitation therapy but without satisfactory improvement.

Exclusion Criteria:

1. Inability to follow instructions.
2. Any visible abnormalities on the hard palate that prevent use of the palatal device.
3. Any mental or physical illness beyond the secondary effects of vestibular loss that prevent recognition or effective use of the alternative feedback.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui Tang, Ph.D, Study Director — Innervo Technology LLC
Locations (2):
- United States (2):
  - MU ENT Hearing and Balance Center, Columbia, Missouri
  - Blue Ridge Physical Therapy, Independence, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Participants' age and history of illness (i.e., vestibular loss) will be shared. However, no personal identifiable information will be collected and shared.

REFERENCES:
- [Background] Tang H, Beebe DJ. An oral tactile interface for blind navigation. IEEE Trans Neural Syst Rehabil Eng. 2006 Mar;14(1):116-23. doi: 10.1109/TNSRE.2005.862696. PMID 16562639
- [Background] Tang H; Beebe DJ. Design and microfabrication of a flexible oral electrotactile display. Journal of Microelectromechanical Systems. 2003 Feb;12(1):29-36.
- [Background] Danilov YP, Tyler ME, Skinner KL, Hogle RA, Bach-y-Rita P. Efficacy of electrotactile vestibular substitution in patients with peripheral and central vestibular loss. J Vestib Res. 2007;17(2-3):119-30. PMID 18413905
- [Background] Dozza M, Horak FB, Chiari L. Auditory biofeedback substitutes for loss of sensory information in maintaining stance. Exp Brain Res. 2007 Mar;178(1):37-48. doi: 10.1007/s00221-006-0709-y. Epub 2006 Oct 5. PMID 17021893
- [Background] Wall C 3rd, Merfeld DM, Rauch SD, Black FO. Vestibular prostheses: the engineering and biomedical issues. J Vestib Res. 2002-2003;12(2-3):95-113. PMID 12867668
- [Background] Brown KE, Whitney SL, Wrisley DM, Furman JM. Physical therapy outcomes for persons with bilateral vestibular loss. Laryngoscope. 2001 Oct;111(10):1812-7. doi: 10.1097/00005537-200110000-00027. PMID 11801950
- [Background] Agrawal Y, Carey JP, Della Santina CC, Schubert MC, Minor LB. Disorders of balance and vestibular function in US adults: data from the National Health and Nutrition Examination Survey, 2001-2004. Arch Intern Med. 2009 May 25;169(10):938-44. doi: 10.1001/archinternmed.2009.66. PMID 19468085
- See also: Vestibular Disorder-Overview — https://vestibular.org/sites/default/files/page_files/Vestibular%20Disorders%20an%20Overview.pdf
- See also: The Human Balance System — https://vestibular.org/sites/default/files/page_files/Human%20Balance%20System.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single group, recruited at MU balance clinic
Pre-assignment Details: Patient with full denture was excluded
Groups:
- Patients Diagnosed With Vestibular Dysfunction: Subjects with vestibular deficiency will try the intraoral electronic balance aid to see whether there is improvement in balance.
  EquiCue (Intraoral Electronic Balance Aid): When the device is worn, a subject will receive small electrical pulses on roof of the mouth as alternative feedback of head tilting or movement.
Period: Overall Study
Arm/Group | Patients Diagnosed With Vestibular Dysfunction
Started | 4
Completed | 3
Not Completed | 1
Not completed — No symptoms in clinic/personal leave | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients Diagnosed With Vestibular Dysfunction
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Equilibrium Score
Description: Equilibrium scores for each trial for each condition from Sensory Organization Test (EquiTest). Conditions: 1-6; with or without using EquiCue intraoral balance aid. Equilibrium scores were generated from the EquiTest CDP (computerized dynamic posturography) platform to assess standing balance of a patient ranging from 0 (all falls) to 100 (perfect balance with no sway), with higher scores indicating better balance performance. An equilibrium score of 70 and above is considered normal.
Time Frame: July 2016 - October 2016 (~ 4 months)
Population: One patient did not have any symptoms during clinical visits, and she did not finish the three test sessions for balance and DGI. Her results were excluded for comparison. The remaining participants included one male and two females.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Diagnosed With Vestibular Dysfunction
Number analyzed (Participants) | 3
score on a scale
  Equilibrium score without device | 63 (4.97)
  Equilibrium with device | 69.67 (9.88)

2. Secondary Outcome: Perceived Intensity Level
Description: The perceived Intensity level (from 0 to 5) as judged by a patient in response to pulsed stimuli applied on the palatal surface after adjustment of device settings for that patient. 1 - barely perceptible, 2 - weak, 3 - good, 4 - strong, 5 - painful.
Time Frame: July 2016 - October 2016 (~ 4 months)
Population: Even though 1 patient did not show any symptoms during clinical visits, all 4 patients each had a device custom made and tested for perceived intensity levels.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Diagnosed With Vestibular Dysfunction
Number analyzed (Participants) | 4
units on a scale | 2.91 (0.12)

3. Secondary Outcome: Dynamic Gait Index
Description: A subject's gait is evaluated by a physical therapist when no device is worn and when alternative sensory feedback of head movement is presented to the patient using the device. 7 walking exercises were administrated for each DGI test, with a score in the range of 0 - 3 (0 for severely impaired and 3 for normal gait) for each exercise, and a total score in the range of 0 - 21 for each test.
Time Frame: July 2016 - October 2016 (~ 4 months)
Population: One patient did not show any symptoms during clinical visits, and her DGIs were excluded for comparison.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Diagnosed With Vestibular Dysfunction
Number analyzed (Participants) | 3
score on a scale
  DGI score without device | 17.22 (2.80)
  DGI score with device | 19.11 (3.00)

4. Secondary Outcome: Analog Visual Scale for the Perceived Frequency of Stimulation Pulses
Description: A patient's assessment of the speed of pulses to quantify perceptual difference in the pulse frequencies of the feedback on the palatal surface.
Time Frame: July 2016 - October 2016 (~ 4 months)
Population: This test process was not performed for patients with vestibular dysfunction as it is such a tedious process that it is not practical for a patient with dizziness to complete.
Arm/Group | Patients Diagnosed With Vestibular Dysfunction
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: July 2016 - October 2016 (~ 4 months)
Arm/Group | Patients Diagnosed With Vestibular Dysfunction
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No